CLINICAL TRIAL: NCT01815112
Title: Benefit of MRI and 18F-FDG PET Imaging in the Early Diagnosis of Alzheimer-like Dementia
Brief Title: Early Diagnosis of Alzheimer-like Dementia: Benefit of MRI and PET Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative re-organization of the department. Referent physician left the hospital.
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI07-PR-MEYER1; 2007-A01009-44 (Registry Identifier: RCB)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Vascular Dementia
Keywords: Neurodegenerative disease; Elderly; Dementia; FDG-PET; MRI; Neuroimaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia, Vascular; Neurodegenerative Diseases; Dementia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Alzheimer (Experimental): Alzheimer patients detected via conventional clinical and neuropsychological tests. They will undergo Magnetic resonance imaging and positron emission tomography examinations.
  Interventions: Other: Magnetic resonance imaging; Other: Positron emission tomography
- Vascular dementia (Experimental): Vascular dementia patients detected via conventional clinical and neuropsychological tests. They will undergo magnetic resonance imaging and positron emission tomography examinations.
  Interventions: Other: Magnetic resonance imaging; Other: Positron emission tomography
- Mild cognitive impairment (MCI) (Experimental): Mild cognitive impairment (MCI) patients detected via conventional clinical and neuropsychological tests. They will undergo magnetic resonance imaging and positron emission tomography examinations.
  Interventions: Other: Magnetic resonance imaging; Other: Positron emission tomography
- Healthy subjects (MRI) (Experimental): Healthy subjects agreeing to undergo magnetic resonance imaging examination.
  Interventions: Other: Magnetic resonance imaging
- Healthy subjects (PET) (Experimental): Cognitively healthy subjects. These subjects are people addressed in the nuclear medicine department for cancer-related positron emission tomography examination. If they agree, an extended neuropsychological test will assess that they do not suffer any cognitive disorder.
  Interventions: Other: Positron emission tomography

INTERVENTIONS:
Other: Magnetic resonance imaging — CSF flow measurement at Sylvius' aqueduct and cervical levels. Apparent diffusion coefficient and fractional anisotropy determination in corpus callosum, cingulum and hippocampus.
  Other Names: Flow MRI; Brain MRI; Diffusion weighted imaging
  Arms: Alzheimer; Healthy subjects (MRI); Mild cognitive impairment (MCI); Vascular dementia
Other: Positron emission tomography — Tissue-time activity curves in hippocampus, cingulum, medio-temporal cortex and choroid plexus.
  Other Names: Dynamic PET imaging
  Arms: Alzheimer; Healthy subjects (PET); Mild cognitive impairment (MCI); Vascular dementia

SUMMARY:
The physio-pathology of Alzheimer's disease (AD) remains unknown and there is no cure. Thus, the search for objective markers of preclinical first signs of cognitive impairment, is currently a major public health issue. Early detection of the disease is a major challenge to hope to slow or even stop the neurodegenerative process before the stage of dementia.

In AD the investigators observe:

* A reduction in the volume of brain hippocampi associated with an alteration of the diffusion of water molecules in the white matter.
* A structural brain degeneration coupled with a decrease in cerebral glucose metabolism.

Recent publications show that cerebrospinal fluid (CSF)flow is also altered, probably due to dysfunction of the choroid plexus. Hence the potential interest to study is, in addition to conventional imaging, the imaging of CSF dynamics and choroid plexus metabolism. In that aim,the investigators use two imaging modalities:

* Magnetic resonance imaging (MRI) is used to assess blood and CSF flow in the brain
* Positron emission tomography (PET) is used to assess glucose metabolism in grey/white matter and also in choroid plexus.

The investigators expect that, because of choroid plexus atrophy in AD, CSF flow would be altered as well as glucose metabolism dynamic in choroid plexus.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 65
* Participants (or representatives) gave their written informed consent
* Dementia diagnosed according to Diagnostic and Statistical Manual of Mental Disorders (DSM IV) criteria
* For Alzheimer arm: probable Alzheimer based disease according to NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association ) criteria
* For vascular dementia: diagnosis based on NINDS-AIREN (National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherche et l'Enseignement en Neurosciences) criteria
* For MCI: diagnosis based on Petersen index

Exclusion Criteria:

* Claustrophobia
* Diabetes
* Cardiovascular disease
* Glycemia over 1.3 g/L
* Lumbar puncture within one week before MRI examination
* Non MR-compatible implant
* Suspected brain metastases
* No informed consent signature

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Dynamic FDG (fluoro-deoxyglucose) PET | Day 2
  Extraction of tissue time-activity curves ; notably in choroid plexus.

SECONDARY OUTCOMES:
Aqueductal CSF flow | Day 1
  Measurement of CSF flow at the Sylvius' aqueduct level. Calculation of the corresponding stroke volume.
Follow-up MRI | Day 365
  MRI examination of MCI patients after one year in order to assess CSF flow differences in MCI how converted to Alzheimer.
Follow-up PET | Day 366
  Dynamic FDG PET examination of MCI patients after one year in order to assess FDG dynamic evolution in MCI how converted to Alzheimer.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Etienne MEYER, MD,PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Rouen, Rouen, Haute Normandie
  - CHU Amiens, Amiens, Picardie